CLINICAL TRIAL: NCT04351685
Title: A Multicenter, Phase III, Double-blind, Randomized, Active-controlled Study to Evaluate the Efficacy and Safety of VPM1002 in Comparison to BCG in Prevention of Mycobacterium Tuberculosis Infection in Newborn Infants
Brief Title: Evaluation of Efficacy and Safety of VPM1002 in Comparison to BCG in Prevention of Tb Infection in Infants
Acronym: VPM1002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: Serum Life Science Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VPM1002-MN-3.05TB
Record Dates: First submitted 2020-04-01; First posted 2020-04-17 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Mycobacterium Tuberculosis Infection
Keywords: Bacterial and fungal diseases
MeSH Terms: conditions — Tuberculosis; Mycoses | interventions — VPM1002 recombinant BCG vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is designed as a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VPM1002 (Experimental): Total 3470 subjects will be enrolled in VPM1002 arm.
  Single dose of VPM1002 will be administered.
  Interventions: Biological: VPM1002
- BCG SII (Active Comparator): Total 3470 subjects will be enrolled in BCG SII arm.
  Single dose of BCG SII will be administered.
  Interventions: Biological: BCG SII

INTERVENTIONS:
Biological: VPM1002 — The active ingredient of the recombinant BCG vaccine, VPM1002 is Mycobacterium bovis A dose of 0.05 ml will be administered intradermally.
  Manufactured by the Serum Institute of India Pvt. Ltd., India
  Diluent: 1 ml of Water for injection/vial
  Arms: VPM1002
Biological: BCG SII — Commercially available BCG vaccine from Serum Institute of India Pvt. Ltd. A dose of 0.05 ml will be administered intradermally.
  Manufactured by the Serum Institute of India Pvt. Ltd., India
  Diluent: 1 ml of Sodium Chloride for injection/vial Injection
  Arms: BCG SII

SUMMARY:
The trial is designed as a phase III, double-blind, multicenter, randomized, single administration, active-controlled, parallel-group design with two groups of newborn infants receiving either VPM1002 or BCG SII (1:1 allocation) to assess the efficacy, safety and immunogenicity of VPM1002 against Mtb infection.

DETAILED DESCRIPTION:
The trial is designed as a phase III, double-blind, multicenter, randomized, single administration, active-controlled, parallel-group design with two groups of newborn infants receiving either VPM1002 or BCG SII (1:1 allocation) to assess the efficacy, safety and immunogenicity of VPM1002 against Mtb infection.

Healthy male or female newborn infants will be centrally randomized to receive the allocated vaccine, stratified by the HIV status of the mother. Single dose of VPM1002 or BCG SII will be administered (within 14 days of birth) strictly intradermally.

ELIGIBILITY:
Inclusion Criteria:

A Maternal

1. Age: 18 years or older at screening.
2. Willing to comply with the trial protocol, available and willing to allow her child to complete all the trial assessments and must have signed an Informed Consent form that has been approved by respective Site Ethics Committee.
3. No symptoms or signs of active TB at the time of participant's enrolment.
4. Parent / guardian who intends to remain in the trial area with the child should be reachable by phone during the trial period.
5. For HIV-unexposed group: Test negative for HIV within two months prior to the newborn infant's vaccination. Test result must be documented, in absence of which a HIV test must be performed at the infant screening visit.
6. For the HIV-exposed group: Test positive for HIV and test result must be documented. If documentation is missing, a HIV test must be performed at the screening visit. The newborn infant's mother must have enrolled for standard antiretroviral therapy (ART) at least 2 months before the participant's birth
7. No participation in an interventional clinical trial within 3 months prior to the participant's birth. In addition, if mother is breast-feeding then she must not participate in another clinical trial during the current trial period while breastfeeding.

B Infant

1. Healthy male or female newborn infant.
2. Birth weight of at least 2,300 g.
3. Test negative for HIV by PCR at screening if born to an HIV-infected mother.
4. No participation in an interventional clinical trial prior to enrolment. Participant should not take part in another clinical trial for the duration of the current trial period.

Exclusion Criteria:

A Maternal

1. Any reported or suspected substance abuse during pregnancy.
2. House-hold contact with active TB (defined as residing in the same house as an individual with active TB) within the 3 months prior to enrolment.

B Infant

1. Fever at the time of enrolment.
2. Eczema or other significant skin lesion or infection at the site/s of injection as per protocol.
3. Receipt of routine BCG vaccine (as per vaccination record).
4. Clinically suspected sepsis.
5. Clinically suspected sepsis.
6. Any malignant condition.
7. Any clinically significant severe congenital malformation, which may interfere with the evaluation of the safety, efficacy or immunogenicity of the vaccine.
8. Concomitant treatment with medication that may significantly affect immune function (e.g. systemic corticoids, immunosuppressive drugs) before trial vaccination. (Note: Routine medication given at birth such as topical antibiotics for eye care and vitamins A and K are permitted. In HIV-exposed newborn infants prevention of mother-to-child transmission (PMTCT) based on standard of care is allowed, but must be documented.)
9. Receipt of blood products or immunoglobulin before trial vaccination.

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6940 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Incident cases of QFT conversion, indicating Mtb infection | Minimum of 12 months and maximum of 36 months

SECONDARY OUTCOMES:
The rate of TB disease in children receiving VPM1002 compared to BCG SII. Incident cases of sustained QFT conversion, indicating sustained Mtb infection. | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Prasad Kulkarni, MD, Study Director — Serum Institute of India Pvt. Ltd.
Locations (12):
- Centre de Recherches Médicales de Lambaréné, Lambaréné, Gabon
- Kenya (2):
  - Kenya Medical Research Institute / Center for Respiratory Disease Research, Nairobi
  - Kenya Medical Research Institute - Center for Respiratory Disease Research, Siaya
- South Africa (5):
  - Empilweni Services and Research Unit (ESRU), Johannesburg, Coronation Ville
  - Family Center for Research with Ubuntu, Cape Town
  - Mecru Clinical Research Unit, Medunsa
  - Respiratory and Meningeal Pathogens Research Unit, Soweto
  - South African Tuberculosis Vaccine Initiative, Worcester
- Tanzania (2):
  - The national institute for Medical Research (NIMR) - Mbeya Medical Research Center (MMRC), Mbeya, Mbeya
  - Ifakara Health Institute, Dar es Salaam
- Uganda (2):
  - Medical Research Council / Uganda Virus Research Institute and London School of Hygiene and Tropical Medicines (MRC/UVRI and LSHTM) Uganda Research Unit, Entebbe
  - Makerere University/CISMAC, Kampala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giersing B, Mo AX, Hwang A, Baqar S, Earle K, Ford A, Deal C, Dull P, Friede M, Hall BF. Meeting summary: Global vaccine and immunization research forum, 2023. Vaccine. 2025 Feb 6;46:126686. doi: 10.1016/j.vaccine.2024.126686. Epub 2025 Jan 5. PMID 39752894